CLINICAL TRIAL: NCT06453837
Title: Double Blinded Randomized Placebo Controlled Clinical Study for the Evaluation of the Efficacy of One Active Ingredient Incorporated Into a Food Supplement
Brief Title: Clinical Study for the Efficacy Evaluation of a Food Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mibelle Group Biochemistry (Industry)
Collaborators: Inovapotek, Pharmaceutical Research And Development Lda (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CIP no. P016C23 (v01)
Record Dates: First submitted 2024-01-23; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Spot Pigmented; Wrinkle
Keywords: Food Supplement; Apple mint extract; Skin spots; Depigmenting effect; Skin tone evenness; Skin whitening/brightening; Skin hydration; Skin firmness; Skin radiance
MeSH Terms: conditions — Exanthema

STUDY DESIGN:
Intervention Model Description: The subjects are randomly divided in two groups, the test group, taking the active ingredient (Mentha Suaveolens extract) incorporated into a food supplement and the placebo group, taking the food supplement without the active ingredient. Each subject is randomly assigned to one of the groups (Group I or Group II) according to a Table of Random Numbers created on Microsoft Office Excel.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigational and comparator products are alphabetically coded, using the codes A and B, by inovapotek's personnel not involved in the clinical study in order for the study to be performed in a double blinded fashion.
  Subjects and Investigators enrolled in this study will not know to what product each code corresponds. The traceability of the products during and after the clinical investigation will be achieved by assignment of a code number and a batch number to each product.
  Each subject is randomly assigned to one of the groups (Group I or Group II) according to a Table of Random Numbers created on Microsoft Office Excel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active ingredient incorporated into a food supplement (Experimental): The investigational product (Ref.: S-1171b) is packed on a 200ml bottle and each bottle have 50 capsules of food supplement, manufactured by Mibelle Biochemistry (Bolimattstr. 1, CH - 5033 Buchs).
  Each subject of this group takes 1 capsule of the food supplement per day, with lunch, for 84 consecutive days.
  Interventions: Other: Mentha Suaveolens extract incorporated into a food supplement
- Placebo product (Placebo Comparator): The comparator product is a placebo (Ref.: S-1171a) with the same formulation as the investigational product, except for the active ingredient, on a 200ml bottle and each bottle have 50 capsules of food supplement, manufactured by Mibelle Biochemistry (Bolimattstr. 1, CH - 5033 Buchs).
  Each subject of this group takes 1 capsule of comparator product per day, with lunch, for 84 consecutive days.
  Interventions: Other: Placebo product

INTERVENTIONS:
Other: Mentha Suaveolens extract incorporated into a food supplement — Each subject of this group takes 1 capsule of the food supplement per day, with lunch, for 84 consecutive days.
  Arms: Active ingredient incorporated into a food supplement
Other: Placebo product — Each subject of this group takes 1 capsule of comparator product per day, with lunch, for 84 consecutive days.
  Arms: Placebo product

SUMMARY:
The primary aim of this in vivo clinical study is to evaluate the depigmenting effect of an active ingredient incorporated into a food supplement through the evaluation of the melanin variation parameter, assessed with the equipment Antera 3D (Miravex, Ireland), after 28 consecutive days of food supplement's once-daily intake, in comparison with the baseline and a placebo.

The secondary objective of this study is to evaluate in vivo the depigmenting effect of the same active ingredient incorporated into a food supplement through the evaluation of the melanin variation parameter, assessed with the equipment Antera 3D (Miravex, Ireland), after 56 and 84 consecutive days of food supplement's once-daily intake.

Other goals of this clinical study are to evaluate in vivo the effect of the same active ingredient incorporated into a food supplement, after 28, 56 and 84 consecutive days of a once-daily intake, in comparison with the baseline and a placebo (1) on skin whitening/brightening through the evaluation of the L* parameter, assessed with the equipment Antera 3D (Miravex, Ireland), (2) on the skin colour homogeneity through the measurement of the ITAº (Individual Typology Angle) parameter, assessed with the equipment Colorimeter® CL400, (3) on the skin tone evenness through the measurement of the standard deviation of the skin colour, assessed with the equipment Colorimeter® CL400, (4) on the skin density of the dermis, measured with the equipment Episcan 35 MHz (Longport Inc, United States), (5) on skin hydration assessed through capacitance measurements with the equipment Corneometer® CM825, (6) on the skin firmness, skin overall elasticity and skin total deformation measured with the equipment Cutometer® SEM 575 (Courage+Khazaka electronic GmbH, Germany), and (7) on skin radiance through clinical evaluation performed by an expert.

It is also objective of this clinical study to evaluate (8) subjects' tolerance, acceptability, perception of efficacy and future use/purchase intention towards the food supplements by filling out a subjective evaluation questionnaire after 28, 56 and 84 consecutive days of food supplement's once-daily intake.

DETAILED DESCRIPTION:
The primary aim of this in vivo clinical study is to evaluate the depigmenting effect of an active ingredient incorporated into a food supplement through the evaluation of the melanin variation parameter, assessed with the equipment Antera 3D (Miravex, Ireland), after 28 consecutive days of food supplement's once-daily intake, in comparison with the baseline and a placebo.

The secondary objective of this study is to evaluate in vivo the depigmenting effect of the same active ingredient incorporated into a food supplement through the evaluation of the melanin variation parameter, assessed with the equipment Antera 3D (Miravex, Ireland), after 56 and 84 consecutive days of food supplement's once-daily intake.

Other goals of this clinical study are to evaluate in vivo the effect of the same active ingredient incorporated into a food supplement, after 28, 56 and 84 consecutive days of a once-daily intake, in comparison with the baseline and a placebo (1) on skin whitening/brightening through the evaluation of the L* parameter, assessed with the equipment Antera 3D (Miravex, Ireland), (2) on the skin colour homogeneity through the measurement of the ITAº (Individual Typology Angle) parameter, assessed with the equipment Colorimeter® CL400, (3) on the skin tone evenness through the measurement of the standard deviation of the skin colour, assessed with the equipment Colorimeter® CL400, (4) on the skin density of the dermis, measured with the equipment Episcan 35 MHz (Longport Inc, United States), (5) on skin hydration assessed through capacitance measurements with the equipment Corneometer® CM825, (6) on the skin firmness, skin overall elasticity and skin total deformation measured with the equipment Cutometer® SEM 575 (Courage+Khazaka electronic GmbH, Germany), and (7) on skin radiance through clinical evaluation performed by an expert.

It is also objective of this clinical study to evaluate (8) subjects' tolerance, acceptability, perception of efficacy and future use/purchase intention towards the food supplements by filling out a subjective evaluation questionnaire after 28, 56 and 84 consecutive days of food supplement's once-daily intake.

In order to perform this study, 110 female healthy subjects, with ages between 25 and 60 years old, presenting mild to moderate fine lines and wrinkles, mild to moderate skin spots and phototype III to V, according to the Fitzpatrick phototyping scale, are enrolled. The subjects are randomly divided in two groups, the test group, taking the active ingredient incorporated into a food supplement and the placebo group, taking the food supplement without the active ingredient.

A 2 weeks washout period is performed, if subject has taken any kind of supplements (Vitamins, antioxidants, nutraceuticals) before the beginning of the study. In this period subjects cannot use any kind of supplements.

Each subject shall take 1 capsule of the food supplement per day, with lunch, for 84 consecutive days.

ELIGIBILITY:
Inclusion criteria for Group I/II:

* Gender: Female;
* Age: between 25 and 60 years old;
* Having signed an Informed Consent Form (ICF);
* Willingness, ability and likeliness to comply with all the study procedures and restrictions;
* Available during the entire study period;
* Understanding Portuguese language: Portuguese-speaking subjects capable of reading the documents;
* Presenting skin phototype between III to V according to the Fitzpatrick phototyping scale;
* Presenting mild to moderate fine lines and wrinkles on the crow's feet area on at least one side of the face;
* Presenting mild to moderate skin spots on the forehead and/or cheek of at least one side of the face;
* Presenting self-perceived normal do dry skin type;
* Having a stable means of contraception for at least 3 months before beginning of the study and not changing the means of contraception during the study;
* Willing to not use any other products/treatments/home remedies except the provided products and their normal make-up and cleansing products during the study;
* Willing to not expose excessively to sunlight (sun exposure not more than one hour daily and during that time use of umbrella to cover face), and to not attend artificial sun beds during the study;
* Willingness to apply sunscreen 15-30 minutes before sun exposure and to record its use in the daily log;

Exclusion criteria for Group I/II:

* Known allergy or known history of hypersensitivity to the components of the investigational and comparative products (e.g. mint-based products), to bar cleansing products, cosmetics, creams/lotions, artificial jewellery or anything else;
* Currently participating in a clinical study that may interfere with the present study or having participated in a clinical study with face products or food supplements for less than 1 month before the beginning the study;
* Having any history of significant, acute, or chronic dermatological conditions or diseases (e.g. eczema, psoriasis, sclerosis, acne condition, skin allergies etc.);
* Having any history of systemic diseases or even infections (e.g. diabetes, hypertension, cardiovascular, upper respiratory infections, urinary tract infections etc.);
* Presenting signs or symptoms of irritated or damaged facial skin (any skin area which shows any desquamation, severe dryness, skin picking, etc.);
* Having performed major anti-ageing, anti-wrinkles, rejuvenating, whitening, depigmenting and smoothing treatments on the 30 days preceding the beginning of the study (including but not limited to: topical hydroquinone, topical treatments with benzoyl peroxide, retinoid, face lifts, cryotherapy, injectable fillers, electrosurgery, CO2 laser, peelings, laser or intense pulsed light) or with intention to perform it during the study;
* Having performed pharmacological treatments systemic/topical on the 30 days before the beginning of the study or currently taking medication that may impair the study;
* Having changed the usual daily cosmetic products (including cleansing and make-up products) and/or habits in the face on the 15 days preceding the beginning of the study;
* Intention of prolonged solar exposure or going to tanning beds on the 15 days preceding the beginning of the study and/or during the course of the study
* Having an activity-based outdoor occupation or with hobbies requiring excessive sun exposure;
* Smokers or users of tobacco products, including vaping products;
* Having history of heavy caffeine consumption of ≥ 4 cups in a day;
* Having high-risk drinking as defined by consumption of 4 or more alcohol containing beverages on any day or 8 or more alcohol containing beverages per week.
* Pregnancy or intention to conceive during the study;
* Breast-feeding.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Skin depigmenting evaluation | From enrollment to the end of treatment: before (t0) and after 28 (t1), 56 (t2) and 84 (t3) consecutive days of food supplement's once-daily intake.
  The skin depigmenting is evaluated by measuring the melanin variation parameter with the equipment Antera 3D before (t0) and after 28 (t1), 56 (t2) and 84 (t3) consecutive days of a once-daily intake, in comparison with the baseline and a placebo.
  Variation of melanin provides information on the uniformity of the pigment. The variation is inversely proportional to the uniformity of the pigment, meaning that a lower melanin variation corresponds to a higher degree of uniformity, consequently a decrease on the melanin variation parameter means that the skin tone is more even.
Skin whitening/brightening evaluation | From enrollment to the end of treatment: before (t0) and after 28 (t1), 56 (t2) and 84 (t3) consecutive days of food supplement's once-daily intake.
  The skin whitening/brightening is evaluated by measuring the L*parameter, with the equipment Antera 3D before (t0) and after 28 (t1), 56 (t2) and 84 (t3) consecutive days of a once-daily intake, in comparison with the baseline and a placebo.
  The skin whitening/brightening evaluation depigmenting translated in the L* parameter represents lightness from black to white on a scale of 0 to 100. The higher the value of the L* parameter, the lighter the skin colour, which represents a whitening effect.

OTHER OUTCOMES:
Skin colour and skin tone evenness evaluation | From enrollment to the end of treatment: before (t0) and after 28 (t1), 56 (t2) and 84 (t3) consecutive days of food supplement's once-daily intake.
  The colour of the skin of each subject is evaluated by measuring the ITAº and the homogeneity of the skin tone by measuring the standard deviation of skin colour with equipment Colorimeter® CL400 before (t0) and after 28 (t1), 56 (t2) and 84 (t3) consecutive days of food supplement's once-daily intake.
  A higher ITA value means a lighter skin tone and, consequently, an increase of the ITA parameter represents a lightening effect.
Skin density evaluation of the dermis | From enrollment to the end of treatment: before (t0) and after 28 (t1), 56 (t2) and 84 (t3) consecutive days of food supplement's once-daily intake.
  High resolution ultrasound images are taken on the cheekbone of the opposite hemiface of each subject with the equipment Episcan 20 MHz (Longport Inc, United States) before (t0) and after 28 (t1), 56 (t2) and 84 (t3) consecutive days of food supplement's once-daily intake. Measurements of the skin density of the dermis of the taken images of the cheekbone are performed, calculating the mean value of 9 determinations per image.
  Greater density (refers to the increase in the amount of cellular tissue underlying the skin's surface) provides structural support and reduces the appearance of wrinkles and sagging. Skin that has lost its density has likely been experiencing signs of a breakdown in collagen, elastin, and overall skin structure resulting in sagging, fine lines and wrinkles. So, an increase in the density of the dermis is related to an improvement of the skin quality.
Skin hydration evaluation | From enrollment to the end of treatment: before (t0) and after 28 (t1), 56 (t2) and 84 (t3) consecutive days of food supplement's once-daily intake.
  Skin capacitance is assessed instrumentally on the opposite hemiface of each subject on the forehead with the equipment Corneometer® CM825 (Courage+Khazaka electronic GmbH, Germany), before (t0) and after 28 (t1), 56 (t2) and 84 (t3) consecutive days of food supplement's once-daily intake, by applying slight pressure.
  An increase of the obtained values indicates an improvement of the skin hydration and, consequently, a hydrating effect of the product.
Skin firmness evaluation | From enrollment to the end of treatment: before (t0) and after 28 (t1), 56 (t2) and 84 (t3) consecutive days of food supplement's once-daily intake.
  The skin firmness (R7; Ur/Uf) is evaluated by the suction method with the equipment Cutometer® on the randomized hemiface of each subject (along the zygomatic bone) before(t0) and after 28(t1), 56(t2) and 84(t3) consecutive days of food supplement's once-daily intake.
  Regarding this parameter, a higher R7 value means an increase on the skin recuperation capacity after deformation and, consequently, on the skin firmness. It must increase and be closer to 1 with the improvement of the skin.
Skin overall elasticity evaluation | From enrollment to the end of treatment: before (t0) and after 28 (t1), 56 (t2) and 84 (t3) consecutive days of food supplement's once-daily intake.
  The skin overall elasticity (R2; Ua/Uf), is evaluated by the suction method with the equipment Cutometer® on the randomized hemiface of each subject (along the zygomatic bone) before(t0) and after 28(t1), 56(t2) and 84(t3) consecutive days of food supplement's once-daily intake.
  Regarding this parameter, a higher R2 value means an increase on the viscoelastic recuperation index and, consequently, on the skin overall elasticity. It must increase and be closer to 1 with the improvement of the skin.
Skin total deformation evaluation | From enrollment to the end of treatment: before (t0) and after 28 (t1), 56 (t2) and 84 (t3) consecutive days of food supplement's once-daily intake.
  The skin total deformation (R0; Uf), is evaluated by the suction method with the equipment Cutometer® on the randomized hemiface of each subject (along the zygomatic bone) before(t0) and after 28(t1), 56(t2) and 84(t3) consecutive days of food supplement's once-daily intake.
  Regarding this parameter, a lower Uf value means a decrease on the R0 parameter and, consequently, on the total elastic and plastic deformation of the skin. If the total deformation of the skin decreases, it may indicate an improvement in skin elasticity.
Clinical evaluation of skin radiance | From enrollment to the end of treatment: before (t0) and after 28 (t1), 56 (t2) and 84 (t3) consecutive days of food supplement's once-daily intake.
  The clinical assessment of skin radiance is performed by an expert, on the face of each subject, under standardized light and position conditions, before (t0) and after 28 (t1), 56 (t2) and 84 (t3) consecutive days of food supplement's once-daily intake.
  For the radiance evaluation according to the Griffith's scale, a decrease on the rating score is related to an increase on the category, which means an improvement on the radiance parameter.
Subjective evaluation questionnaire | From enrollment to the end of treatment: after 28 (t1), 56 (t2) and 84 (t3) consecutive days of food supplement's once-daily intake.
  A subjective evaluation questionnaire is performed to evaluate the tolerance, acceptability, efficacy, future use and purchase intention towards the investigational product and the comparator product Placebo, after 28 (t1), 56 (t2) and 84 (t3) consecutive days of food supplement's once-daily intake.
Daily Log Questionnaire Analysis | From enrollment to the end of treatment: sence day 1 (t0) to 84 (t3) consecutive days of food supplement's once-daily intake.
  Subjects fill in a subject diary (daily log) during the course of the study to record: Products usage, Adverse events, Concomitant medication, Sunscreen usage, Make-up usage, Compliance with other inclusion or exclusion criteria.
Photographs | From enrollment to the end of treatment: before (t0) and after 28 (t1), 56 (t2) and 84 (t3) consecutive days of food supplement's once-daily intake.
  Photographs of the face (frontal and profile views) are taken with the equipment Visia-CR (Canfield Scientific Europe, Netherlands), before (t0) and after 28 (t1), 56 (t2) and 84 (t3) consecutive days of food supplement's once-daily intake. Standardized images are captured in the 5 Standard Lighting modes: standard 1, standard 2, cross-polarized, polarized and UV (blue filter) with the measurement room light on.
  Images of 2 selected subjects (one per each product used) are included in the final report and the complete album of photographs is provided to the sponsor at the end of the study.
  The images are used only for qualitative evaluation and client marketing purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Ferreira, Principal Investigator — Inovapotek, Pharmaceutical Research And Development Lda
Locations (1):
- Inovapotek, Pharmaceutical Research And Development Lda, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No
The results will be published in a scientific journal and it is therefore preferable not to give access to the data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT06453837/Prot_SAP_000.pdf